CLINICAL TRIAL: NCT00550433
Title: An Open-Label, Single-Dose, Randomized, 4-Period, Crossover, Bioequivalence Study of Clinical and Commercial Formulations of Bazedoxifene/Conjugated Estrogens in Healthy Postmenopausal Women
Brief Title: Study Evaluating Bazedoxifene/CE in Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3115A1-1117
Record Dates: First submitted 2007-10-25; First posted 2007-10-29 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Postmenopause

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Bazedoxifene/Conjugated Estrogens

SUMMARY:
The purpose of this clinical trial is to study the blood levels of a drug (conjugated estrogens) in the body from one dosage form compared to another. The four formulations of the study drug that eligible participants will receive will contain the same amounts of the same medications. In addition, information will also be obtained regarding the safety and tolerability of the formulations given to healthy postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged 35 to 70 years.
* Spontaneous or surgical amenorrhea for at least 6 months.
* Body mass index (BMI) in the range of 18.0 to 35.0 kg/m2 and body weight greater than or equal to 50 kg.

Exclusion Criteria:

* Hypertension or elevated supine blood pressure (>139 mm Hg systolic or >89 mm Hg diastolic).
* History of any clinically important drug allergy.
* Use of any prescription or investigational drug within 30 days before test article administration.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2007-09; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The plasma concentration data and pharmacokinetic (PK) parameters of BZA and CE.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer